CLINICAL TRIAL: NCT05254535
Title: I-TRUST: Implementation of Teleophthalmology in Rural Health Systems Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-1474; UG1EY032446 (NIH); Protocol Version 1/25/2022 (Other: UW Madison); A536000 (Other: UW Madison); 2022-0121 (Other: UW Certified Not Human Subjects Research)
Record Dates: First submitted 2022-02-23; First posted 2022-02-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Retinopathy
Keywords: Rural Health; Screening; Teleophthalmology; Telemedicine; Preventative Medicine
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Deoxyribonucleases, Type I Site-Specific

STUDY DESIGN:
Intervention Model Description: Cluster-randomized trial with a stepped-wedge initiation of the intervention at each site
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Up to 10 rural health systems will be participating in I-SITE implementation with cluster-randomization of the order of initiation for the intervention. All sites will receive usual care teleophthalmology prior to I-SITE implementation.
  Interventions: Other: I-SITE

INTERVENTIONS:
Other: I-SITE — I-SITE includes coaching facilitation, technical assistance, and an online toolkit to allow primary care clinics to tailor the integration of teleophthalmology into their daily workflows based on each clinic's unique needs and resources. The program includes a series of coaching sessions between a skilled practice facilitator and clinical personnel at each health system.
  Other Names: Implementation for Sustained Impact in Teleophthalmology

SUMMARY:
This pragmatic clinical trial is being conducted to test the effectiveness of I-SITE (Implementation for Sustained Impact in Teleophthalmology), an implementation program to sustain increased diabetic eye screening rates using teleophthalmology in rural, multi-payer health systems. Up to 10 rural health systems providing teleophthalmology to 10,000 patients with diabetes and 100 clinical care personnel participating in the I-SITE intervention will be enrolled for up to 48 months.

DETAILED DESCRIPTION:
The investigators' long-term goal is to reduce vision loss nationwide through widespread teleophthalmology use. The next step in the project is to determine whether I-SITE is an effective, generalizable strategy across multiple rural health systems.

The investigators will test the primary hypothesis that I-SITE will sustain significant diabetic eye screening rate increases of ≥ 20% (e.g., from 40% to ≥ 60%) compared to baseline. The primary outcome measure will be the change in diabetic eye screening rates between baseline and 24 months after initiation of I-SITE implementation. Secondary outcome measures include characterizing pre/post changes in screening rates at 12, 36, and up to 48 months after I-SITE implementation at all sites, follow-up rates for in-person eye care among screen positives, identifying key factors and core implementation components distinguishing high and low teleophthalmology-use health systems following I-SITE implementation, and measuring implementation costs.

I-Site implementation will include:

* Teleophthalmology in primary care clinic
* I-SITE online toolkit
* Technical assistance from study team via email
* Introductory live webinar with question & answer session (30 min) between I-SITE Coach and primary care clinic
* Series of 2 in-person meetings over 6 weeks (45-60 min.) between I-SITE Coach and local implementation team
* Series of 10 monthly teleconferences (15-30 min.) between I-SITE Coach and local implementation team
* Series of 4 quarterly group teleconferences (45-60 min.) between I-SITE Coach and local implementation teams

Aim 1: To test the effectiveness of I-SITE vs. usual care teleophthalmology for increasing diabetic eye screening rates among 10 rural health systems across 6 states. The investigators will use a cluster-randomized study design with a stepped wedge initiation of the intervention to optimize longitudinal assessment of sustained increases in diabetic eye screening rates up to 48 months. The investigators will also measure follow-up rates for in-person eye care among screen positives every 6 months.

Aim 2: To identify key factors and core implementation components that distinguish high and low teleophthalmology-use rural health systems after I-SITE implementation. The investigators will use an explanatory mixed methods design, including interviews with clinicians and health system personnel, to identify workflow strategies, organizational factors, and implementation components that determine the effectiveness of I-SITE implementation.

Aim 3: To determine implementation costs of I-SITE. The investigators will measure implementation costs from a health system perspective, including health system personnel time tracked using structured activity logs.

ELIGIBILITY:
Inclusion Criteria:

* Health system serves rural patients as defined as those patients living in counties considered rural by the federal Office of Management and Budget (OMB)
* Health system has an active clinical teleophthalmology program providing diabetic eye screening in primary care prior to study randomization
* Health system agrees to share de-identified patient data at the requested time intervals

Exclusion Criteria:

* Health system does not serve a rural patient population
* Health system has a diabetic eye screening rate of greater than 50% (e.g., above the national average) as it may limit the ability to measure improvement from I-SITE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Who Complete Annual Diabetic Eye Screening | 24 months
  Comparison of proportion of patients with diabetes adherent with yearly diabetic eye screening guidelines (i.e., "screening rates") between baseline and 24 months following initiation of I-SITE implementation at each site.

SECONDARY OUTCOMES:
Change in Proportion of Patients Who Complete Annual Diabetic Eye Screening | baseline, 12 months, 36 months, 48 months
  Comparison of proportion of patients with diabetes adherent with yearly diabetic eye screening guidelines (i.e., "screening rates") between baseline and 12, 36, and up to 48 months following initiation of I-SITE implementation at each site.
Change in follow-up rates for in-person eye care among screen positive patients | baseline, 12 months, 36 months, 48 months
  Comparison of follow-up rates for in-person eye care among screen positives between baseline and 12, 24, 36, and up to 48 months following initiation of I-SITE implementation at each site.
Identification of workflow strategies, organizational factors, and implementation components that distinguish between health systems with high and low teleophthalmology use | up to 13 months
  An explanatory mixed methods design including interviews and direct observation as data sources will be used. Qualitative interviews with key clinical informants and direct observation of I-SITE Coach and local implementation team meetings are planned. Configurational Comparative Methods (CCM) will combine qualitative data with quantitative data on teleophthalmology use to characterize differences between health systems.
  Key clinical informant interviews will be conducted 1 month prior to and 12 months following initiation of I-SITE implementation. Verbatim transcripts of audio recordings from individual interviews will be coded and analyzed using directed content analysis based on the i-PARiHS framework.
  Qualitative data from fidelity checklists obtained through direct observation of meetings will be coded using a similar analytic approach to that used in the interviews.
  High and low teleophthalmology use will be defined based on the last 6 months of I-SITE implementation.
Mean Implementation Cost | up to 48 months
  Implementation costs determined by structured activity logs and project records of all communications between I-SITE Coach, clinical personnel, and research team.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Liu, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested from other researchers up to 7 years after the completion of the primary outcome by contacting Dr. Yao Liu, the Principal Investigator of this study.
Supporting Information: Study Protocol, SAP
Time Frame: up to 7 years after the completion of the primary outcome

REFERENCES:
- [Background] Liu Y, Carlson JN, Torres Diaz A, Lock LJ, Zupan NJ, Molfenter TD, Mahoney JE, Palta M, Boss D, Bjelland TD, Smith MA. Sustaining Gains in Diabetic Eye Screening: Outcomes from a Stakeholder-Based Implementation Program for Teleophthalmology in Primary Care. Telemed J E Health. 2021 Sep;27(9):1021-1028. doi: 10.1089/tmj.2020.0270. Epub 2020 Nov 19. PMID 33216697
- [Background] Torres Diaz A, Lock LJ, Molfenter TD, Mahoney JE, Boss D, Bjelland TD, Liu Y. Implementation for Sustained Impact in Teleophthalmology (I-SITE): applying the NIATx Model for tailored implementation of diabetic retinopathy screening in primary care. Implement Sci Commun. 2021 Jul 6;2(1):74. doi: 10.1186/s43058-021-00175-0. PMID 34229748
- See also: I-SITE free online toolkit — https://www.hipxchange.org/I-SITE